CLINICAL TRIAL: NCT07068282
Title: Vitamin D3, Mouthwash, Saliva Testing, Covid-19, Antiviral Testing
Brief Title: The Effect of Novel D3 Use as a Mouthwash in COVID-19 Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Sarah Feteih, Consultant, Periodontist, King Faisal Specialist Hospital & Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-32
Record Dates: First submitted 2025-06-24; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2024-01

CONDITIONS: Corona Virus Disease 19 (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- D3 mouthwash in COVID-19 saliva (Experimental)
  Interventions: Drug: Cholecalciferol (vitaminD3)

INTERVENTIONS:
Drug: Cholecalciferol (vitaminD3) — Vitamin D3 mouthwash was prepared for COVID-19 participants, to compare between the saliva only (control group), and with the use of mouthwash in saliva after the participants swish for 60 seconds (experimental group) and compare the effect of vitamin D over the virus in saliva, from both groups by testing via RAT and R-PCR.

SUMMARY:
The PI's goal of this [interventional/clinical trial] is to [explore the antiviral properties of vitamin D3 on saliva samples collected before and after the use of a vitamin D3 mouthwash] in [ adult participants, both genders, with COVID-19 who tested positive on a swab test]. The main question[s] aims to answer [is]:

[Assess the antiviral potential of a novel vitamin D-based mouthwash in COVID-19-positive participants].

PI will compare both [Control group: saliva only- before use of mouthwash], and the [study group: after use of the mouthwash in saliva] to see if there is [any veridical effect present in saliva after running lab tests].

Participants will [self-collect saliva in a given tube (color coded orange), then 10-15 minutes later or more, participants will swish with D3 mouthwash, and will give another sample [saliva + mouthwash] in another (green labeled tube). For each participant, each of the following will be given:

* 2 collecting tubes: orange labeled tube (for saliva collection only) and green labeled tube (for saliva collection after mouthwash use).
* The vial containing vitamin D3 mouthwash.

DETAILED DESCRIPTION:
Twenty-five adult participants confirmed COVID-19-positive, via rapid antigen testing (RAT) thru nasal swabs (NS), followed by saliva samples collected before and after using a vitamin D3 mouthwash. Samples were analyzed using RAT and rapid polymerase chain reaction (R-PCR) to measure viral load.

ELIGIBILITY:
Inclusion criteria:

* Adult participants confirmed positive for COVID-19 by RAT.
* Participants at the King Faisal Specialist Hospital & Research Center in Jeddah (KFSHRC, J) outpatient departments (OPD) and/or department of emergency medicine (DEM).

Exclusion criteria:

* Immunocompromised and/or pregnant participants.
* Pediatric participants and patients aged <18 years.
* Participants on a high-dose vitamin D prescription (i.e., 10, 000 IU or more).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
No effect of D3 mouthwash on saliva of COVID-19 patients | 30-60 minutes was the time frame for each participant, during same day of COVID-19 testing.
  Post-rinse, RAT positivity dropped by 68%, likely due to physical dilution rather than antiviral action. R-PCR showed no significant reduction in viral RNA; in some cases, a slight increase was observed, potentially reflecting a cellular response to D3

CONTACTS AND LOCATIONS:
Locations (1):
- KingFaisal, Jeddah, Saudi Arabia